CLINICAL TRIAL: NCT06791915
Title: The Effect of Mechanical Ventilation on Radiofrequency Ablation in The Treatment of Atrial Fibrillation.
Brief Title: Effect of Mechanical Ventilation on Radiofrequency Ablation in Atrial Fibrillation
Status: Recruiting | Type: Observational
Sponsor: Kocaeli City Hospital (Other Government)
Responsible Party: Principal Investigator, Merve Yazici Kara, Principal Investigator, Kocaeli City Hospital
Other Study IDs: 2024-149
Record Dates: First submitted 2025-01-07; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Radiofrequency Ablation; Atrial Fibrillation; Mechanical Ventilation
Keywords: Atrial Fibrillation; Ablation; general anesthesia
MeSH Terms: conditions — Atrial Fibrillation | interventions — Radiofrequency Ablation; Famciclovir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Flow Controlled Mechanical Ventilation (FCV): Controlled ventilation parameters and hemodynamic and respiratory values (systolic pressure, diastolic pressure, peak heart rate, peripheral oxygen saturation, fraction of inspired oxygen (FiO2)), and Bispectral Index monitoring (BIS) values in the patient's preferred FCV mode will be recorded. Ablation lesion parameters including mean ablation time per lesion, mean contact force, mean impedance drop, mean ablation index, and procedural characteristics including total procedure time, total ablation time, and total RF time will also be recorded. Clinical outcomes, including freedom from all atrial arrhythmias and short and long-term procedural complications, will also be recorded at routine patient follow-up.
  Interventions: Procedure: Radiofrequency Ablation with FCV.
- Volume Controlled Mechanical Ventilation (VCV): Controlled ventilation parameters and hemodynamic and respiratory values (systolic pressure, diastolic pressure, peak heart rate, peripheral oxygen saturation, fraction of inspired oxygen (FiO2)), and Bispectral Index monitoring (BIS) values in the patient's preferred VCV mode will be recorded. Ablation lesion parameters including mean ablation time per lesion, mean contact force, mean impedance drop, mean ablation index, and procedural characteristics including total procedure time, total ablation time, and total RF time will also be recorded. Clinical outcomes, including freedom from all atrial arrhythmias and short and long-term procedural complications, will also be recorded at routine patient follow-up.
  Interventions: Procedure: Radiofrequency Ablation with VCV.

INTERVENTIONS:
Procedure: Radiofrequency Ablation with FCV. — Treatment of atrial fibrillation patients with radiofrequency ablation under general anesthesia with Flow Controlled Mechanical Ventilation (FCV).
  Groups: Flow Controlled Mechanical Ventilation (FCV)
Procedure: Radiofrequency Ablation with VCV. — Treatment of atrial fibrillation patients with radiofrequency ablation under general anesthesia with Volume Controlled Mechanical Ventilation (VCV).
  Groups: Volume Controlled Mechanical Ventilation (VCV)

SUMMARY:
Radiofrequency ablation (RFA) for atrial fibrillation (AF) is performed under general anesthesia. The success of the procedure depends on the safe contact of the catheter electrode with the myocardium. Movement of the catheter tip due to respiratory changes can result in inadequate lesion formation and AF recurrence.

The success of AF ablation depends on the adequacy of energy delivered to the myocardium and the durability of pulmonary vein isolation (PVI). Poor energy delivery and tissue heating during ablation are a major cause of procedural failure in RFA. To improve the success of the PVI procedure, efforts are underway to optimize catheter stability and contact force. However, catheter force and stability are influenced by respiration-induced thoracic motion, highlighting the importance of controlled breathing for further optimization. Fluoroscopy and ablation times during electroanatomic mapping-guided AF ablations improved with controlled mechanical ventilation. General anesthesia improved catheter contact.

Low tidal volume, high respiratory rate (FCV), pressure controlled mechanical ventilation (PCV), volume controlled mechanical ventilation (VCV), pressure controlled volume assured mechanical ventilation (PRVC) can be used in investigators' hospital. The literature offers no definitive proof that one ablation procedure is superior to another.

DETAILED DESCRIPTION:
Radiofrequency ablation for the treatment of atrial fibrillation (AF) has recently been performed under general anesthesia with patients connected to a mechanical ventilator device. There are studies showing that whether patients are connected to spontaneous or controlled ventilation directly affects the results of the ablation procedure. In the ablation procedure, safe myocardial tissue contact of the catheter electrode determines predictable lesion size distribution and ultimately procedural success. Therefore, contact force has been a reliable marker in predicting the ability to deliver an effective transmural lesion. Catheter tip movement due to respiratory changes may lead to inadequate lesion formation, potentially resulting in AF recurrence. In the existing literature, high-frequency jet ventilation (HFJV) has been reported to increase catheter stability, improve tissue contact and reduce AF recurrence due to reduced thoracic motion. An alternative strategy was used by simulating very low tidal volume ventilation with high respiratory rate with a flow similar to HFJV with standard anesthesia devices.

The incidence of atrial fibrillation recurrence following catheter ablation depends on various patient-level factors and procedural techniques. An important determinant of success in AF ablation is the adequacy of the energy delivered to the cardiac tissue and the durability of pulmonary vein isolation (PVI). Approximately 20% of patients undergoing AF ablation require re-ablation within 12 months, regardless of technique. AF recurrence following ablation occurs mainly through pulmonary vein electrical reconnection, and the rate of ≥ 1 reconnected pulmonary vein during AF reablation is >80%. Inadequate energy delivery and tissue heating due to insufficient contact or challenging anatomical locations during ablation is one of the main culprits of procedure failure in radiofrequency ablation (RFA). Therefore, efforts to improve the success of the PVI procedure include optimizing catheter stability and contact force. Thus, catheter force and stability are highly influenced by respiratory-induced thoracic movement, demonstrating the importance of controlled breathing for further ablation optimization. Fluoroscopy and ablation times during electroanatomic mapping-guided AF ablations have improved significantly with the use of controlled mechanical ventilation. To improve catheter contact, general anesthesia with controlled breathing has been used for better procedural success than conscious sedation.

To date, there are no randomized clinical trials in the literature demonstrating the superiority of one mode of ventilation over another during the ablation procedure. Low tidal volume, high respiratory rate (FCV, Flow Controlled Ventilation), pressure controlled mechanical ventilation (PCV), volume controlled mechanical ventilation (VCV), pressure controlled volume guaranteed mechanical ventilation (PRVC) can be applied with the mechanical ventilator equipment available in the anesthesiology and reanimation clinic of investigators' hospital. However, HFJV mechanical ventilator mode cannot be applied in general anesthesia patients in accordance with the facilities of investigators' hospital. In addition, there is no definite information in the literature about the superiority of any mode over the other for ablation procedure. Therefore, different mechanical ventilation modes are applied in ablation procedures in investigators' hospital according to the preferences of the practitioner. Investigators believe that there is a need for studies on the modes used in ablation procedures performed under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with atrial fibrillation
* planned to receive radiofrequency ablation treatment under general anesthesia
* all patients over 18 years of age

Exclusion Criteria:

- Patients undergoing ablation under sedation and/or local anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All ASA I-II-III patients over 18 years of age with a diagnosis of atrial fibrillation who were planned to receive radiofrequency ablation treatment under general anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Radiofrequency ablation procedure duration. | At the end of the ablation procedure (Ablation time varies between 1 and 3 hours)
  The effect of mechanical ventilation mode during radiofrequency ablation procedure on procedure duration.
Change From Baseline Electrocardiography After Radiofrequency Ablation. | At the end of the ablation procedure (Ablation time varies between 1 and 3 hours)
  Change in baseline ECG during radiofrequency ablation procedure showing the effect of mechanical ventilation mode on procedural success.
After radiofrequency ablation procedure atrial fibrillation recurrence rate. | In one month after procedure.
  The effect of mechanical ventilation mode during radiofrequency ablation procedure on atrial fibrillation recurrence rate.

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli City Hospital, Kocaeli, Turkey (Türkiye)